CLINICAL TRIAL: NCT06206772
Title: The Role of Resting State Networks Connectivity in Cluster Headache: a HD-EEG Study
Brief Title: Resting State Functional Connectivity in Cluster Headache
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: HD-EEG in Cluster Headache
Record Dates: First submitted 2023-12-15; First posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Cluster Headache; Headache Disorders
MeSH Terms: conditions — Cluster Headache; Headache Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy subjects
  Interventions: Diagnostic Test: Resting state HD-EEG recording
- Episodic cluster headache, active
  Interventions: Diagnostic Test: Resting state HD-EEG recording
- Episodic cluster headache, remission
  Interventions: Diagnostic Test: Resting state HD-EEG recording
- Chronic cluster headache
  Interventions: Diagnostic Test: Resting state HD-EEG recording

INTERVENTIONS:
Diagnostic Test: Resting state HD-EEG recording — All subjects will be recorded with a resting state HD-EEG recording. 12 minutes in the eyes closed and 12 minutes in the eyes open condition.

SUMMARY:
Cluster headache is a highly disabling primary headache disorder, characterized by severe, excruciating, recurrent unilateral headache attacks. Typically, attacks' onset displays a circadian rhythm, and bout recurrence happens in a circannual fashion. Notably, the mechanisms underlying the shift between the remission phase and cluster bout are poorly understood.

Thus, the investigators aim to study brain connectivity in episodic cluster headache patients. Additionally, an explorative analysis of functional connectivity in chronic cluster headache patients will be performed.

DETAILED DESCRIPTION:
Electroencephalogram (EEG) is widely available as a powerful mean to non-invasively study brain connectivity. High density EEG (HD-EEG), enables to record electrical brain activity with high temporal and spatial resolution. Through the analysis of brain oscillations across different frequency bands (from alpha to delta), it can evaluate sensory, pain processing and information integration, thus detecting potential markers or predictors for therapeutic interventions.

Previous neurophysiological studies focused on EEG and to assess functional connectivity or spectral analysis in migraine patients, with no data in cluster headache. Conventional studies found higher slow wave activity (predominantly theta) in the inter-ictal phase and higher excitability in the visual cortex during visual aura.

In 2016 a resting state study showed a predominance of low frequency bands in the ictal phase. The interictal and ictal phases patients also presented a diffuse lower coherence, suggesting low functional connectivity. Furthermore, an altered spatial connectivity for lower alpha-band activities was found in the interictal phases during sensory stimulation by means of HD-EEG, suggesting a thalamocortical dysrhythmia.

The primary aim of the study is to evaluate changes in functional connectivity in episodic cluster headache patients, comparing the active phase with the remission phase. Additionally, an explorative analysis of functional connectivity in chronic cluster headache patients will be performed.

Study design:

Episodic cluster headache patients (eCH) will be evaluated in two separate timepoints: during the active phase (T0), defined as at least one week of active bout, and in remission phase (T1), defined as at leat 14 days without headache and without any ongoing preventive medication. During each visit, clinical data will be collected, and an HD-EEG will be performed.

Chronic cluster headache patients (cCH) will be evaluated in a single timepoint, and healthy controls will undergo HD-EEG registration once.

HD-EEG registration:

Participants will perform 4 recordings (6 minutes each) in resting-state condition, 2 with opened eyes, and 2 with closed eyes, in a randomized order.

The investigators will analyze the resting state FC among six resting state networks (Default mode network, Dorsal attention network, Ventral attention network, Language network , Somatomotor network and Visual network) in the following frequency bands: alfa 8-12 Hz, beta 13-30 Hz, gamma 31-80 Hz, theta 4-7 Hz. delta 1-3 Hz.

Acquisition parameters will be: High-Pass: 0.5 Hz; Low-Pass: 100 Hz; Notch: 50 Hz. For analysis of HD-EEG data, a tailored analysis pipe-line that was previously developed and validated to reconstruct neural sources from cortical/subcortical gray matter will be performed. EEG signals will be band-pass filtered (1-80 Hz) and down-sampled at 250 Hz. Biological artifacts will be rejected using Independent Component Analysis (ICA). EEG signals will be referenced with a customized version of the Reference Electrode Standardization Technique (REST). A matrix will estimate the relationship between the measured scalp potentials and the dipoles corresponding to brain sources. Sources reconstruction will be performed with the exact low-resolution brain electromagnetic tomography (eLORETA) algorithm

Statistical plan:

The sample size was computed with the freeware online platform www.openepi.com. As there are no previous studies on HD-EEG functional connectivity in cluster headache, our sample size analysis was based on the work of Bjork (Bjork et al., 2009). A difference between groups in the theta relative power band equal to 0.04 (±0.04) will be considered as clinically meaningful. Considering a two-tailed t-test for the comparison with confidence interval 95%; power: 80%, the minimum suggested sample size was 20 subjects for group.

A preliminary normality analysis will be performed to decide whether to use parametric or non-parametric methods, through Shapiro Wilk test.

Numerical variables will be described as mean and standard deviation (or median and quartiles if appropriate), categorical variables as raw numbers and percentages.

Functional connectivity analyses will be conducted for separate bands and eyes closed registration.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of 3.1.1 episodic cluster headache, or 3.1.2 chronic cluster headache, according to the International Classification of Headache Disorders-3 (ICHD-3) criteria
* History of at least 1 year of disease
* For the active-phase recording (T0) in eCH, no preventive medication ongoing or verapamil at a stable dose for at least 2 weeks
* For the remission-phase recording (T1), no preventive medication ongoing, and at least 14 headache-free days since preventive discontinuation

Exclusion Criteria:

* Previous or actual history of epilepsy
* Diagnosis of dementia o mental retardation
* Diagnosis of psychiatric illness according to Diagnostic and Statistical Manual of Mental Disorders V
* Other concomitant type of headache (except for sporadic tension type headache)
* Chronic pain conditions
* Pregnancy or breastfeeding
* Concomitant use of electrical stimulators, pace-makers, metallic clips or other metallic foreign bodies
* Previous head surgery
* Ongoing neuroactive prevention therapies or other drugs, or psychoactive substances possibly interfering with EEG recording (eg benzodiazepines)
* Other conditions possibly influencing EEG recording
* Brain anomalies detected on MRI

Healthy controls (HCs)

Inclusion Criteria:

* Age and sex-matched healthy volunteers, without history of headache disorders except sporadic tension-type headache according to ICHD-3 criteria

Exclusion Criteria:

* Previous or actual history of epilepsy
* Diagnosis of dementia o mental retardation
* Diagnosis of psychiatric illness according to Diagnostic and Statistical Manual of Mental Disorders V
* Chronic pain conditions
* Pregnancy or breastfeeding
* Concomitant use of electrical stimulators, pace-makers, metallic clips or other metallic foreign bodies
* Previous head surgery
* Ongoing neuroactive prevention therapies or other drugs, or psychoactive substances possibly interfering with EEG recording (eg benzodiazepines)
* Other conditions possibly influencing EEG recording

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with episodic and chronic cluster headache patients attending the outpatient clinic of the Headache Science & Neurorehabilitation Center of the IRCCS Mondino Foundation (Pavia, Italy).
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Difference in absolute functional connectivity values (continuous variable, without unit of measurement) in resting state networks (RSN-FC) in episodic cluster headache patients between active and remission phases | Through study completion, an average of 2 years
  To compare HD-EEG functional connectivity in episodic cluster headache patients between the two phases of the disease
Differences in absolute functional connectivity values (continuous variable, without unit of measurement) in resting state networks (RSN-FC) between episodic cluster headache patients and healthy controls | Through study completion, an average of 2 years
  To compare HD-EEG functional connectivity between episodic cluster headache patients in the two phases of the disease and healthy controls

SECONDARY OUTCOMES:
Differences in absolute functional connectivity values (continuous variable, without unit of measurement) in resting state networks (RSN-FC) between episodic cluster headache patients and chronic cluster headache patients | Through study completion, an average of 1 year
  To compare HD-EEG functional connectivity between episodic cluster headache patients and chronic cluster headache patients
Differences in absolute functional connectivity values (continuous variable, without unit of measurement) in resting state networks (RSN-FC) between chronic cluster headache patients and healthy controls | Single evaluation in chronic cluster headache (cCH) vs. healthy controls (HCs)
  To compare HD-EEG functional connectivity between chronic cluster headache patients and healthy controls

OTHER OUTCOMES:
To assess for correlations between clinical features of episodic cluster headache and absolute functional connectivity values in resting state networks (RSN-FC) | Through study completion, an average of 2 years
  To search for correlations between clinical variables and HD-EEG functional connectivity in episodic cluster headache

CONTACTS AND LOCATIONS:
Overall Officials: Roberto De Icco, MD, Principal Investigator — Headache Science ahd Neurorehabilitation Research Center
Locations (1):
- Headache Science & Neurorehabilitation Center, Pavia, Italy

REFERENCES:
- [Background] Headache Classification Committee of the International Headache Society (IHS) The International Classification of Headache Disorders, 3rd edition. Cephalalgia. 2018 Jan;38(1):1-211. doi: 10.1177/0333102417738202. No abstract available. PMID 29368949
- [Background] Bjork MH, Stovner LJ, Engstrom M, Stjern M, Hagen K, Sand T. Interictal quantitative EEG in migraine: a blinded controlled study. J Headache Pain. 2009 Oct;10(5):331-9. doi: 10.1007/s10194-009-0140-4. Epub 2009 Aug 25. PMID 19705061
- [Background] Coppola G, Di Lorenzo C, Parisi V, Lisicki M, Serrao M, Pierelli F. Clinical neurophysiology of migraine with aura. J Headache Pain. 2019 Apr 29;20(1):42. doi: 10.1186/s10194-019-0997-9. PMID 31035929
- [Background] de Tommaso M, Trotta G, Vecchio E, Ricci K, Siugzdaite R, Stramaglia S. Brain networking analysis in migraine with and without aura. J Headache Pain. 2017 Sep 29;18(1):98. doi: 10.1186/s10194-017-0803-5. PMID 28963615
- [Background] Cao Z, Lin CT, Chuang CH, Lai KL, Yang AC, Fuh JL, Wang SJ. Resting-state EEG power and coherence vary between migraine phases. J Headache Pain. 2016 Dec;17(1):102. doi: 10.1186/s10194-016-0697-7. Epub 2016 Nov 2. PMID 27807767
- [Background] Chamanzar A, Haigh SM, Grover P, Behrmann M. Abnormalities in cortical pattern of coherence in migraine detected using ultra high-density EEG. Brain Commun. 2021 Apr 2;3(2):fcab061. doi: 10.1093/braincomms/fcab061. eCollection 2021. PMID 34258580
- [Background] Semprini M, Bonassi G, Barban F, Pelosin E, Iandolo R, Chiappalone M, Mantini D, Avanzino L. Modulation of neural oscillations during working memory update, maintenance, and readout: An hdEEG study. Hum Brain Mapp. 2021 Mar;42(4):1153-1166. doi: 10.1002/hbm.25283. Epub 2020 Nov 17. PMID 33200500
- [Background] Aoki Y, Ishii R, Pascual-Marqui RD, Canuet L, Ikeda S, Hata M, Imajo K, Matsuzaki H, Musha T, Asada T, Iwase M, Takeda M. Detection of EEG-resting state independent networks by eLORETA-ICA method. Front Hum Neurosci. 2015 Feb 10;9:31. doi: 10.3389/fnhum.2015.00031. eCollection 2015. PMID 25713521